CLINICAL TRIAL: NCT04949659
Title: Postoperative Pain in Children After Low-Pressure Versus Medium-Pressure Pneumoperitoneum in Laparoscopic Surgery
Brief Title: Low vs Medium Pressure Pneumoperitoneum
Acronym: LoMePneu
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1001
Record Dates: First submitted 2021-06-21; First posted 2021-07-02 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Appendicitis Acute
Keywords: Pneumoperitoneum; Pressure; Pain
MeSH Terms: conditions — Appendicitis; Pneumoperitoneum; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low pressure pneumoperitoneum (Experimental): Use of low pressure pneumoperitoneum during laparoscopic appendectomy
  Interventions: Procedure: Laparoscopic appendectomy
- Medium pressure pneumoperitoneum (Experimental): Use of medium pressure pneumoperitoneum during laparoscopic appendectomy
  Interventions: Procedure: Laparoscopic appendectomy

INTERVENTIONS:
Procedure: Laparoscopic appendectomy — Laparoscopic appendectomy performed with defined, randomized to level of pressure for pneumoperitoneum

SUMMARY:
The purpose of this study is to asses whether the pressure used for the pneumoperitoneum during laparoscopic surgery in children affects their postoperative pain levels.

ELIGIBILITY:
Inclusion Criteria:

* Prepped and consented for diagnostic laparoscopy for likely acute appendicitis
* 5 years or older
* 15 kg or more
* Parents/legal custodian give consent, patient shows no signs of unwillingness to participate
* Patient is hemodynamically stable

Exclusion Criteria:

* Clinical signs of four quadrant peritonitis as a clinical sign of perforated appendicitis
* Suspected perityphlitic abscess on preoperative ultrasound
* Preexisting conditions making postoperative assessment of extent of pain and its localization very difficult or impossible, e.g. conditions that are associated with pronounced developmental delays or with communication difficulties
* Parents have inadequate knowledge of German language to understand Informed consent
* Child has inadequate knowledge of German language to allow elicitation of Pain Scores

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2021-09-27 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain score on postoperative day one (abdominal pain) | Postoperative day one.
  Postoperative pain score for abdominal pain on postoperative day one after laparoscopic appendectomy using the Faces Pain Score Revised (FPS-R score), a self-reported pain score using drawn faces with values from 0 (no pain) to 10 (most pain). It is validated for use in studies with children.

SECONDARY OUTCOMES:
Postoperative pain scores during postoperative phase (abdominal pain) | Through study completion, an average of 3 days
  Postoperative pain score for abdominal pain on further postoperative days (excluding day one, which is primary outcome) after laparoscopic appendectomy using the Faces Pain Score Revised (FPS-R score), a self-reported pain score using drawn faces with values from 0 (no pain) to 10 (most pain). It is validated for use in studies with children.
Postoperative pain scores during postoperative phase (shoulder pain) | Through study completion, an average of 3 days
  Postoperative pain score for shoulder pain during hospitalisation after laparoscopic appendectomy using the Faces Pain Score Revised (FPS-R score), a self-reported pain score using drawn faces with values from 0 (no pain) to 10 (most pain). It is validated for use in studies with children.
Length of operation | Intraoperative
  Length of operation in minutes
Length of stay | Through study completion, an average of 3 days
  Length of stay in hospital in hours
Intra- and postoperative complications | Through study completion, an average of 3 days
  Intra- and postoperative complications during hospitalisation
Analgesic use | Through study completion, an average of 3 days
  Number and dose (mg/kg) of standard analgesia, as well as so called "rescue" doses

CONTACTS AND LOCATIONS:
Overall Officials: Hannah R Neeser, MD, Principal Investigator — University Children's Hospital of Zurich
Locations (1):
- University Children's Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gurusamy KS, Vaughan J, Davidson BR. Low pressure versus standard pressure pneumoperitoneum in laparoscopic cholecystectomy. Cochrane Database Syst Rev. 2014 Mar 18;2014(3):CD006930. doi: 10.1002/14651858.CD006930.pub3. PMID 24639018
- [Background] Ozdemir-van Brunschot DM, van Laarhoven KC, Scheffer GJ, Pouwels S, Wever KE, Warle MC. What is the evidence for the use of low-pressure pneumoperitoneum? A systematic review. Surg Endosc. 2016 May;30(5):2049-65. doi: 10.1007/s00464-015-4454-9. Epub 2015 Aug 15. PMID 26275545
- [Background] McGrath PJ, Walco GA, Turk DC, Dworkin RH, Brown MT, Davidson K, Eccleston C, Finley GA, Goldschneider K, Haverkos L, Hertz SH, Ljungman G, Palermo T, Rappaport BA, Rhodes T, Schechter N, Scott J, Sethna N, Svensson OK, Stinson J, von Baeyer CL, Walker L, Weisman S, White RE, Zajicek A, Zeltzer L; PedIMMPACT. Core outcome domains and measures for pediatric acute and chronic/recurrent pain clinical trials: PedIMMPACT recommendations. J Pain. 2008 Sep;9(9):771-83. doi: 10.1016/j.jpain.2008.04.007. Epub 2008 Jun 17. PMID 18562251